CLINICAL TRIAL: NCT04128423
Title: A Phase 1 Dose Escalation With Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMV564 Alone and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: Study of AMV564 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amphivena Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMV564-301
Record Dates: First submitted 2019-10-10; First posted 2019-10-16 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-05

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: immunotherapy; anti-CD33; T-cell engager

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMV564 (Experimental)
  Interventions: Biological: AMV564

INTERVENTIONS:
Biological: AMV564 — AMV564 will be administered daily

SUMMARY:
This Phase 1 study is designed to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of AMV564 alone and in combination with Pembrolizumab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
AMV564-301 is a Phase 1, open-label, multicenter dose-escalation with expansion trial in patients with locally advanced or metastatic solid tumors. In the dose-escalation portion of the study, cohorts of patients will receive AMV564 alone or in combination with Pembrolizumab at increasing dose levels to determine the maximum tolerated dose (MTD) and/or the recommended dose for expansion. In the expansion portion of the study, one or more cohorts of patients will receive AMV564 at the MTD or recommended dose to further evaluate safety, tolerability, and clinical activity.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Histologically or cytologically documented, incurable or metastatic solid tumor that is advanced (non-resectable) or recurrent and progressing since the last anti-tumor therapy and for which no recognized standard therapy exists
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or per other criteria best suited for the specific tumor type being evaluated
* Willing to complete all scheduled visits and assessments at the institution administering therapy

Key Exclusion Criteria:

* Treatment with any local or systemic antineoplastic therapy (including chemotherapy, hormonal therapy, or radiation) within 3 weeks prior to first dose of AMV564
* Major trauma or major surgery within 4 weeks prior to first dose of AMV564
* Prior treatment with chimeric antigen receptor (CAR) T-cell therapy or T-cell engager therapy
* Chronic use of corticosteroids in excess of 10 mg daily of prednisone or equivalent within 4 weeks prior to first dose of AMV564
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1 except for alopecia
* Known, central nervous system (CNS) disease involvement, or prior history of National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Grade ≥ 3 drug-related CNS toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Through study completion, an average of 19 months
  As measured by the incidence, nature and severity of adverse events (AEs) and serious AEs
Maximum tolerated dose of AMV564 in subjects with advanced solid tumors | During Dose Escalation, an average of 6 months
  As determined based on the occurrence of dose-limiting toxicity
Preliminary evaluation of AMV564 efficacy in subjects enrolled in the expansion phase | During Dose Expansion, an average of 1 year
  As measured by the objective response rate (ORR)

SECONDARY OUTCOMES:
Maximum observed drug concentration (Cmax) of AMV564 | Through study completion, an average of 19 months
  Measured by plasma concentration
Concentration at steady state (Css) of AMV564 | Through study completion, an average of 19 months
  Measured by plasma concentration
Time of the maximum drug concentration (Tmax) of AMV564 | Through study completion, an average of 19 months
  Measured by plasma concentration
Apparent terminal half-life (t½) of AMV564 | Through study completion, an average of 19 months
  Measured by plasma concentration
Area under the concentration-time curve (AUC) of AMV564 | Through study completion, an average of 19 months
  Measured by plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chun, MD, Study Director — Amphivena Therapeutics
Locations (11):
- United States (11):
  - UCLA, Los Angeles, California
  - Advent Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No